CLINICAL TRIAL: NCT05720442
Title: Efficacy Assessment of Chinese Herbal Medicine Tangweian Recipe Treating Participants With Diabetic Gastroenteropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jiaxing Tian, Dr., Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFIMD2022B06
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Gastroenteropathy
Keywords: Diabetic Gastroenteropathy
MeSH Terms: interventions — mosapride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tangweian Recipe Group (Experimental): 1. Tangweian formula granule (30g per bag), 1 bag per time, twice a day, take it with warm water after meals.
  2. 1 mosapride citratetablet per time, 3 times a day, take it with meals.
  Interventions: Drug: Tangweian Recipe; Drug: Mosapride Citrate
- Mosapride Citrate Group (Active Comparator): 1 mosapride citratetablet per time, 3 times a day, take it with meals.
  Interventions: Drug: Mosapride Citrate

INTERVENTIONS:
Drug: Tangweian Recipe — The Tangweian recipe is a combination of several Chinese herbs
  Arms: Tangweian Recipe Group
Drug: Mosapride Citrate — The mosapride citrate tablets will be administrated.

SUMMARY:
This study is a randomized, positive drug parallel-controlled clinical trial in participants with diabetic gastroenteropathy. A total of 60 participants will be recruited for the study, all of whom are diagnosed as diabetes mellitus combined with gastroenteropathy. The subjects will be divided randomly into two groups and treated with either Tangweian Recipe+mosapride citrate tablets or mosapride citrate tablets for four weeks. The primary outcome will be the change in gastroparesis symptom severity, as measured by the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptoms Daily diary Index-Daily Diary (ANMS GCSI-DD). And participants will be seen for a clinic evaluation at weeks 0 and 4, during which symptom scores, adverse events and treatment compliance will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years at the time of their consent;
2. Those diagnosed with diabetic gastrointestinal lesions with gastrointestinal symptoms such as nausea/vomiting, early satiety, bloating, and epigastric pain for more than 3 months or longer;
3. History of symptoms of mellitus for at least 5 years leading up to the Screening Visit and Blood glucose stable within 1 month;
4. Mean Gastroparesis Cardinal Symptom Index (GCSI) score ≥ 2; or delayed gastric emptying confirmed at screening by gastric emptying breath test (GEBT);
5. TCM Syndrome differentiation as spleen deficiency and stomach stagnation syndrome;
6. Signed informed consent.

Exclusion Criteria:

1. Patients with diabetic ketoacidosis, hyperosmolar nonketotic diabetic coma, severe infection, and surgery in recent one month;
2. Patients with gastrointestinal reactions caused by glucose-lowering drugs and patients treated with GLP-1 class drugs;
3. Have a history of or are suffering from severe gastrointestinal disease
4. Gastrectomy, fundoplication, vagotomy, pyloroplasty, bariatric surgery, or gastric stimulation device surgically implanted within the last year;
5. Combination of severe cardiovascular and cerebrovascular diseases, hepatic and renal insufficiency, psychiatric patients, drug abuse and dependence;
6. Women who are pregnant, preparing for pregnancy or breastfeeding;
7. Patients who participated in other clinical studies within one month prior to participating in this study or were participating in other clinical studies;
8. According to the judgment of the researcher, other diseases or conditions that reduce the possibility of enrollment or complicate the enrollment, such as frequent changes in working environment and unstable living environment, are likely to cause loss of follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Sub-scores of the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptoms Index-Daily Diary (ANMS GCSI-DD) | Baseline to Week 4
  Change from Baseline at weeks 0 through 4 as measured by patient's daily diary entries during participation in the study.
Patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) | 0 week, 4 weeks

SECONDARY OUTCOMES:
Changes from Baseline Fasting Blood Glucose at 4 weeks | 0 week, 4 weeks
Changes from Baseline Body Mass Index at 4 weeks | 0 week, 4 weeks
Change from Baseline TCM Symptom Score at 4 weeks | 0 week, 4 weeks
SF-36 Health Survey Questionnaire | 0 week, 4 weeks

OTHER OUTCOMES:
Adverse events (AEs) | 0 week, 4 weeks

REFERENCES:
- [Derived] Zhang YX, Yin RY, Zhang YJ, Ji HY, Ma JZ, Zhang C, Zhang LL, Wu XA, Li M, Tian JX. Efficacy and safety of tangweian recipe in the treatment of diabetic gastroparesis: a protocol for a non-inferiority, double-blind, active drug, randomized controlled clinical trial. BMC Complement Med Ther. 2025 Nov 27;26(1):7. doi: 10.1186/s12906-025-05104-5. PMID 41310560